CLINICAL TRIAL: NCT06013774
Title: Interventional X-ray and Scintigraphy Imaging of 99mTc-MAA During the Radioembolisation Pretreatment Procedure
Acronym: IXSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Hugo de Jong, Principal Investigator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NL71365.041.20
Record Dates: First submitted 2023-07-06; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid imaging during the pre-treatment procedure of radioembolization (Experimental): Hybrid imaging will be performed on patients undergoing the pre-treatment procedure of radioembolization
  Interventions: Device: IXSI

INTERVENTIONS:
Device: IXSI — Hybrid imaging with IXSI will be performed during the radioembolization pre-treatment procedure

SUMMARY:
To establish the safety and feasibility of interventional x-ray and scintigraphy imaging during the pre-treatment procedure of hepatic radioembolization

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have given written informed consent and comply with the requirements of the study protocol.
2. Must be aged 18 years or over.
3. Must be selected to undergo a 99mTc-MAA procedure as part of their radioembolisation treatment.
4. Sufficiently fit to undergo an additional examination time of 30-90 minutes.
5. Have a CT acquired less than 6 weeks before the pre-treatment radioembolisation procedure.

Exclusion Criteria:

1. Patients expected to require more than two injection positions for radioembolisation treatment.
2. Pregnancy or nursing.
3. Patients suffering from psychic disorders that make a comprehensive judgement impossible, such as psychosis, hallucinations and/or depression.
4. Patients who are declared incompetent.
5. Previous enrollment in the present study
6. Claustrophobia
7. The last dose of prior chemotherapy has been received less than weeks prior to the planned 99mTc-MAA pre-treatment procedure.
8. Radiation therapy within the last 4 weeks before the planned 99mTc-MAA pre-treatment procedure
9. Major surgery within the last 4 weeks prior to the planned 99mTc-MAA pre-treatment procedure
10. Any unresolved toxicity greater than Common Terminology Criteria for Adverse Events (CTCAE version 5) grade 2 from previous anti-cancer treatment
11. Body weight over 250 kg (because of maximum table load)
12. Patient length over 1.90 m (to fit IXSI geometry)
13. Patient bust line over 135 cm (to fit IXSI geometry)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Device Feasibility | Immediately after surgery
  The feasibility of IXSI will be assessed by questionnaires filled in by interventional radiology personnel

SECONDARY OUTCOMES:
Radioactivity distribution over time | Immediately after surgery
  The radioactivity distribution in the liver segments will be measured over time to assess potential dynamic behavior
Radioactivity distribution in 3D | Immediately after surgery
  The quality of IXSI scans will be assessed by measuring the radioactivity distribution in the liver segments in 3D

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Dietze MMA, Meddens MBM, van Rooij R, Braat AJAT, de Keizer B, Bruijnen RCG, Lam MGEH, Smits MLJ, de Jong HWAM. Safety and Feasibility of Interventional Hybrid Fluoroscopy and Nuclear Imaging in the Work-up Procedure of Hepatic Radioembolization. Radiol Imaging Cancer. 2024 Nov;6(6):e240044. doi: 10.1148/rycan.240044. PMID 39485113